CLINICAL TRIAL: NCT02566187
Title: A Study to Compare the Pharmacokinetics of Fimasartan/Atorvastatin Combination Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FAVC-CT-101
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — fimasartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Subjects of Group 1 take Fimasartan and Atorvastatin Individual Tablets at 1st day as period I. And then, after wash out for 7 days, as period II, subjects of Group 1 take a Fimasartan/Atorvastatin Combination Tablet at 8th day.
  Interventions: Drug: Fimasartan/Atorvastatin Combination Tablet; Drug: Fimasartan; Drug: Atorvastatin
- Group 2 (Other): Subjects of Group 2 take a Fimasartan/Atorvastatin Combination Tablet at 1st day as period I. And then, after wash out for 7 days, as period II, subjects of Group 2 take Fimasartan and Atorvastatin Individual Tablets at 8th day.
  Interventions: Drug: Fimasartan/Atorvastatin Combination Tablet; Drug: Fimasartan; Drug: Atorvastatin

INTERVENTIONS:
Drug: Fimasartan/Atorvastatin Combination Tablet
Drug: Fimasartan
Drug: Atorvastatin

SUMMARY:
A phase I, Open-label, Randomized, Single-dose, 2 x 2 Crossover Study to Compare the Pharmacokinetics of Fimasartan/Atorvastatin Combination Tablet and Coadministration of Fimasartan and Atorvastatin as Individual Tablets in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* a Healthy male subject, aged 19- 50 years

Exclusion Criteria:

* History of clinically significant hypersensitivity to study drug, any other drug
* Hypotension or hypertension
* Active liver disease
* History of gastrointestinal disease
* History of excessive alcohol abuse
* Participation in any other study within 3 months

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration(Cmax) of Fimasartan and Atorvastatin | 0~48 hour after medication
Area under the curve(AUCt) of Fimasartan and Atorvastatin | 0~48 hour after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea